CLINICAL TRIAL: NCT05465421
Title: Clinical and Radiographic Assessment of Buccolingual Bone Dimension Following Socket Preservation With Bone Marrow Mono-nuclear Cell From the Maxillary Tuberosity Combined With Platelet-rich Fibrin Compared With Platelet-rich Fibrin Alone
Brief Title: Effect of Bone Marrow Mononuclear Cell Layer Seeded on Platelet-rich Fibrin on an Alveolar Socket After Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hani Elnahass, clinical professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: cairoU21677
Record Dates: First submitted 2022-06-29; First posted 2022-07-19 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Decayed Teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinding of the participants and the operator is is not applicable, however outcome assessors and biostatistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- socket preservation with platelet rich fibrin PRF alone the implant placement 3 months after (Active Comparator): after extraction socket preservation will be done by using PRF only in the socket and closed the socket by flap advancement.
  Interventions: Other: bone marrow aspiration from maxillary tuberosity and BMMNCs separation to be seeded on PRF and used for socket preservation
- socket preservation with BMMNCs of bone marrow aspirated of maxillary tuberosity (Experimental): after extraction socket preservation will be done by using bone marrow mononuclear cell layer seeded on PRF in the socket and close the socket by flap advancement
  Interventions: Other: bone marrow aspiration from maxillary tuberosity and BMMNCs separation to be seeded on PRF and used for socket preservation

INTERVENTIONS:
Other: bone marrow aspiration from maxillary tuberosity and BMMNCs separation to be seeded on PRF and used for socket preservation — Local anaesthesia will be administered by infiltration or nerve block to achieve the necessary anaesthesia to allow extraction of the indicated tooth Extraction will be done as atraumatically as possible removing any pathosis found that may interfere with bone formation A trapezoidal flap will be created above the extraction socket to allow closure of the surgical site.
  BMMNC will be seeded on platelet rich fibrin and inserted in the socket The flap will be closed by interrupted sutures using 5-0 sutures. implant placement 3 months later

SUMMARY:
Bone marrow aspiration from maxillary tuberosity will be centrifuged to separate the bone marrow mononuclear cell layer using the density gradient separation method, then it will be seeded in a platelet-rich fibrin membrane and used for socket preservation to test the osteogenic ability of the bone marrow mononuclear cell layer in comparison to platelet-rich fibrin alone both ways will receive implant after 3 months

DETAILED DESCRIPTION:
-Research question: In patients with teeth requiring extraction will bone marrow mononuclear cell layer (BMMNC) from maxillary tuberosity seeded on platelet-rich fibrin (PRF) maintain the bucco-palatal/lingual bone dimension during socket preservation compared to platelet rich fibrin alone?

-The rationale for conducting the research: Bone marrow is full of progenitors and cell markers that promote tissue healing. Traditionally bone marrow aspiration is done from extra-oral sites. The obstacle in extra-oral aspiration is the site morbidity and the need to put the patient under general anesthesia.

Intraoral sites like the maxillary tuberosity are filled with marrow spaces that can facilitate the harvesting of marrow cells and reduce the trauma of the harvesting process.

Bone marrow mononuclear cell (BMMNC) transplantation may result in higher rates of bone marrow regeneration in the extraction socket and significantly accelerate bone maturation. It is also suggested that Bone marrow mononuclear cell (BMMNC) plays an important role in bone homeostasis within the extraction socket However, Bone marrow mononuclear cell (BMMNC) has several drawbacks that should be taken into consideration like potential pain during harvest, and variable stem cell quantity and quality depending on age which may hinder the usage of Bone marrow mononuclear cell (BMMNC) in old ages.

The bone regeneration ability of that population of cells and the ease of their acquisition render them good candidates for socket preservation. Hence, the current study aims to evaluate the use of Bone marrow mononuclear cells (BMMNC) obtained from the maxillary tuberosity in promoting bone formation in the alveolar socket after extraction.

-The explanation for the choice of comparators: A parallel group of 12 patients with a non-restorable tooth will undergo extraction and socket preservation.

* In group 1: socket preservation will be done by PRF PRF membrane used in the extraction sockets was demonstrated to promote local soft tissue healing of gums and reduce postoperative pain response. While the effect of PRF to reduce alveolar bone resorption was not significant, PRF was able to increase the quality of the novel bone and enhance the rate of bone formation due to the concentration of growth factors
* In group 2: sock preservation will be done by Bone marrow mononuclear cell (BMMNC) from the maxillary tuberosity on PRF

In the current study, the density gradient separation method technique will be used to harvest BMMNC. This method has been used to enrich the isolated mononuclear cell fraction and has been an essential part of several clinical procedures. The density gradient separation/immediate transplantation method is superior to the in vitro expansion method as the cells are minimally manipulated; there is no invasive enzymatic treatment used. This method allows immediate autologous transplantation of BMAC that minimizes the risk of contamination by decreasing the time of cell handling in cell culture

-Objectives: The objective of the study is to find out the osteogenic potential of BMMNC from the maxillary tuberosity in comparison with PRF alone in socket preservation for delayed implant placement

-Trial design:

The current study will be designed as a:

* Parallel 2 arm
* Randomized Controlled Clinical Trial,
* Allocation ratio 1:1
* Superiority Trial

  * Methods

    . Interventions
  * Preoperative evaluation:
  * Clinical examination & informed consent:

Evaluation of the patient's general condition of the oral cavity, to make sure it complies with the criteria required to be enrolled in the study in terms of oral hygiene, pathological conditions

-Radiographic examination:

Cone beam CT will be taken before proceeding with any procedure to make sure of the restorability of the tooth before extraction, checking for any radiolucency to be removed also to measure bone width before extraction

* Surgical procedures:
* Local anesthesia will be administered by infiltration or nerve block to achieve the necessary anesthesia to allow extraction of the indicated tooth
* Extraction will be done as atraumatically as possible removing any pathosis found that may interfere with bone formation
* Allocation concealment will be broken and socket preservation will be done In group 1
* A trapezoidal flap will be created above the extraction socket to allow closure of the surgical site.
* PRF will be placed in the socket
* The flap will be closed by interrupted sutures using 5-0 sutures. In group 2 (test group)
* A trapezoidal flap will be created above the extraction socket to allow closure of the surgical site.
* BMMNC will be seeded on platelet-rich fibrin and inserted into the socket
* The flap will be closed by interrupted sutures using 5-0 sutures.

BMMNCs aspiration and centrifugation technique:

* Under the supervision of professor: Hani el Nahass and doctor: Omnia k Tawfik A 20 gauge needle will be inserted in the maxillary tuberosity area through the palatal aspect until aspiration is positive
* Aspirate will be collected in a heparin-treated tube (2000:1) using 1ml of anticoagulant citrate dextrose solution (ACD-A) for every 15ml of bone marrow aspiration.
* Aspirate will be centrifuged to separate the BMMNCs using the density gradient separation method.
* Ficoll® Paque Plus (GE Healthcare, Buckinghamshire, UK) bottle will be inverted several times to ensure thorough mixing and 3 ml of the media will be added to a centrifuge tube
* The bone marrow aspirate will be diluted (1:1) with saline and then carefully layered onto the Ficoll gradient and then centrifuged at 2000 rpm for 20 min at room temperature using a multi-speed 4000 rpm vertical rotor.
* The upper layer containing plasma and platelets will be collected using a sterile pipette, leaving the mononuclear cell layer undisturbed at the interface. The layer of mononuclear cells will be transferred to a sterile centrifuge tube using a sterile pipette.
* Postsurgical procedure (three months after socket preservation)
* Local anesthesia will be administered by infiltration or nerve block to achieve the necessary anesthesia
* A flap will be raised at the site of the extracted tooth
* A core biopsy will be harvested by introducing a core drill bit in place of an initial drill
* Sequential drilling will take place to prepare osteotomy to the right size to receive an implant
* Implant will be placed in the osteotomy with the platform flush with the bone
* Flap closure will be achieved by interrupted 5-0 sutures

Histologic processing:

The harvested bone biopsies will be decalcified in ethylene diamine tetra acetic acid (10%) for two weeks. After dehydration in graded series of ethanol, the specimens will be embedded in paraffin and sectioned by a high-speed rotating blade microtome; the sections will be stained with hematoxylin-eosin stain. This will be followed by histomorphometric analysis using the Leica Qwin 500 (Leica microsystems Inc., Switzerland) image analyzer computer system (England). Area percentage (%) of newly formed bone will be calculated

Quantitative real-time polymerase chain reaction (qRT-PCR)

real-time polymerase chain reaction(RT-PCR) will be used to analyze the massenger Ribonucleic acid (mRNA) levels of alkaline phosphatase

• Postoperative instructions and follow-up:

Administration of:

* Antibiotics (Amoxicillin 1g twice daily for 5 days) to prevent any chance of infection. (Eugenio Romeo et al, 2014).
* Anti-inflammatory drugs (NSAIDS; Ibuprofen 600mg three times daily for 5 days) to avoid any chance of edema or pain or swelling
* Antiseptic mouth rinse (0.12% Chlorhexidine oral rinse will be prescribed for 60 seconds two times a day for 14 days.
* The patient will be instructed to follow up for the next 3 months before implant placement

Patient self-care instructions:

* Application of an ice bag to the treated area for the first 24 hours.
* Avoid any brushing and trauma to the surgical site for one week.
* Avoid smoking

  * Outcomes:

PICO:(population-intervention-compatetor-outcome) P: Patients with non-restorable teeth indicated for extraction I: BMMNC from the tuberosity for socket preservation C: Platelet rich fibrin O: Bucco-palatal/lingual bone dimension Prioritization of Outcome Outcome Method of Measurement Unit of Measurement Primary outcome

Secondary objectives To calculate the postoperative pain, patient satisfaction and Alkaline phosphatase measurement in a histological sample of the newly formed bone took 3 months later before implant placement

ELIGIBILITY:
Inclusion Criteria:

* Patients with badly decayed tooth indicated for extraction
* Patients with healthy systemic condition (Medically free)
* Adequate inter-arch space for placement of the implant prosthetic part.
* Good oral hygiene
* Cooperative patients who are willing to commit for 6 months follow up

Exclusion Criteria:

* Smokers
* Pregnant females
* Patient with medical condition that contraindicates surgical procedures
* Patients on medication that may interfere with healing (corticosteroids, bisphosphonate, Chemo/radio therapy).
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as alcoholism or parafunctional habits.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
bucco-palatal width of the alveolar socket after extraction with millimeter by cone-beam computed tomography (CBCT) | 3 months after extraction and socket preservation
  The bucco-palatal width of the alveolar socket after extraction will be measured in millimeter using On Demand software at distinct level (2 , 4, and 6mm from the cerst) at the time of extraction and 3 months later after socket preservation with cone-beam computed tomography (CBCT)

SECONDARY OUTCOMES:
postoperative pain | 14 days
  postoperative pain after the surgery, Visual analogue score from (1 to 10) and 10 is the worst pain
  -A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge

CONTACTS AND LOCATIONS:
Overall Officials: Hani ElNahass, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sauerbier S, Rickert D, Gutwald R, Nagursky H, Oshima T, Xavier SP, Christmann J, Kurz P, Menne D, Vissink A, Raghoebar G, Schmelzeisen R, Wagner W, Koch FP. Bone marrow concentrate and bovine bone mineral for sinus floor augmentation: a controlled, randomized, single-blinded clinical and histological trial--per-protocol analysis. Tissue Eng Part A. 2011 Sep;17(17-18):2187-97. doi: 10.1089/ten.TEA.2010.0516. Epub 2011 Jun 24. PMID 21529247
- [Background] Pasquali PJ, Teixeira ML, de Oliveira TA, de Macedo LG, Aloise AC, Pelegrine AA. Maxillary Sinus Augmentation Combining Bio-Oss with the Bone Marrow Aspirate Concentrate: A Histomorphometric Study in Humans. Int J Biomater. 2015;2015:121286. doi: 10.1155/2015/121286. Epub 2015 Oct 12. PMID 26543482
- [Background] Wildburger A, Payer M, Jakse N, Strunk D, Etchard-Liechtenstein N, Sauerbier S. Impact of autogenous concentrated bone marrow aspirate on bone regeneration after sinus floor augmentation with a bovine bone substitute--a split-mouth pilot study. Clin Oral Implants Res. 2014 Oct;25(10):1175-81. doi: 10.1111/clr.12228. Epub 2013 Jul 22. PMID 23875876
- [Background] Sauerbier S, Stricker A, Kuschnierz J, Buhler F, Oshima T, Xavier SP, Schmelzeisen R, Gutwald R. In vivo comparison of hard tissue regeneration with human mesenchymal stem cells processed with either the FICOLL method or the BMAC method. Tissue Eng Part C Methods. 2010 Apr;16(2):215-23. doi: 10.1089/ten.TEC.2009.0269. PMID 19473102
- [Background] Muschler GF, Boehm C, Easley K. Aspiration to obtain osteoblast progenitor cells from human bone marrow: the influence of aspiration volume. J Bone Joint Surg Am. 1997 Nov;79(11):1699-709. doi: 10.2106/00004623-199711000-00012. PMID 9384430
- [Background] Sununliganon L, Peng L, Singhatanadgit W, Cheung LK. Osteogenic efficacy of bone marrow concentrate in rabbit maxillary sinus grafting. J Craniomaxillofac Surg. 2014 Dec;42(8):1753-65. doi: 10.1016/j.jcms.2014.06.011. Epub 2014 Jun 14. PMID 25052732
- [Background] Duttenhoefer F, Hieber SF, Stricker A, Schmelzeisen R, Gutwald R, Sauerbier S. Follow-up of implant survival comparing ficoll and bone marrow aspirate concentrate methods for hard tissue regeneration with mesenchymal stem cells in humans. Biores Open Access. 2014 Apr 1;3(2):75-6. doi: 10.1089/biores.2014.0003. PMID 24804168
- [Background] de Oliveira TA, Aloise AC, Orosz JE, de Mello E Oliveira R, de Carvalho P, Pelegrine AA. Double Centrifugation Versus Single Centrifugation of Bone Marrow Aspirate Concentrate in Sinus Floor Elevation: A Pilot Study. Int J Oral Maxillofac Implants. 2016 Jan-Feb;31(1):216-22. doi: 10.11607/jomi.4170. PMID 26800181
- [Background] Gapski R, Satheesh K, Cobb CM. Histomorphometric analysis of bone density in the maxillary tuberosity of cadavers: a pilot study. J Periodontol. 2006 Jun;77(6):1085-90. doi: 10.1902/jop.2006.050118. PMID 16734586
- [Background] Al-Ahmady HH, Abd Elazeem AF, Bellah Ahmed NE, Shawkat WM, Elmasry M, Abdelrahman MA, Abderazik MA. Combining autologous bone marrow mononuclear cells seeded on collagen sponge with Nano Hydroxyapatite, and platelet-rich fibrin: Reporting a novel strategy for alveolar cleft bone regeneration. J Craniomaxillofac Surg. 2018 Sep;46(9):1593-1600. doi: 10.1016/j.jcms.2018.05.049. Epub 2018 Jun 2. PMID 30196860
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Zhang Y, Ruan Z, Shen M, Tan L, Huang W, Wang L, Huang Y. Clinical effect of platelet-rich fibrin on the preservation of the alveolar ridge following tooth extraction. Exp Ther Med. 2018 Mar;15(3):2277-2286. doi: 10.3892/etm.2018.5696. Epub 2018 Jan 4. PMID 29456635
- [Background] Mashimo T, Sato Y, Akita D, Toriumi T, Namaki S, Matsuzaki Y, Yonehara Y, Honda M. Bone marrow-derived mesenchymal stem cells enhance bone marrow regeneration in dental extraction sockets. J Oral Sci. 2019;61(2):284-293. doi: 10.2334/josnusd.18-0143. PMID 31217377
- [Background] Marx RE, Tursun R. A qualitative and quantitative analysis of autologous human multipotent adult stem cells derived from three anatomic areas by marrow aspiration: tibia, anterior ilium, and posterior ilium. Int J Oral Maxillofac Implants. 2013 Sep-Oct;28(5):e290-4. doi: 10.11607/jomi.te10. PMID 24066346
- [Background] Iorio-Siciliano V, Blasi A, Nicolo M, Iorio-Siciliano A, Riccitiello F, Ramaglia L. Clinical Outcomes of Socket Preservation Using Bovine-Derived Xenograft Collagen and Collagen Membrane Post-Tooth Extraction: A 6-Month Randomized Controlled Clinical Trial. Int J Periodontics Restorative Dent. 2017 Sep/Oct;37(5):e290-e296. doi: 10.11607/prd.2474. PMID 28817143
- [Background] Barone A, Aldini NN, Fini M, Giardino R, Calvo Guirado JL, Covani U. Xenograft versus extraction alone for ridge preservation after tooth removal: a clinical and histomorphometric study. J Periodontol. 2008 Aug;79(8):1370-7. doi: 10.1902/jop.2008.070628. PMID 18672985
- See also: Bone marrow concentrate and bovine bone mineral for sinus floor augmentation — https://pubmed.ncbi.nlm.nih.gov/21529247/
- See also: Maxillary Sinus Augmentation Combining Bio-Oss with the Bone Marrow Aspirate Concentrate — https://pubmed.ncbi.nlm.nih.gov/26543482/
- See also: Impact of autogenous concentrated bone marrow aspirate on bone regeneration after sinus floor augmentation with a bovine bone substitute — https://pubmed.ncbi.nlm.nih.gov/23875876/
- See also: In vivo comparison of hard tissue regeneration with human mesenchymal stem cells processed with either the FICOLL method or the BMAC method — http://pubmed.ncbi.nlm.nih.gov/19473102/
- See also: Aspiration to obtain osteoblast progenitor cells from human bone marrow: the influence of aspiration volume — http://pubmed.ncbi.nlm.nih.gov/9384430/
- See also: Osteogenic efficacy of bone marrow concentrate in rabbit maxillary sinus grafting — http://pubmed.ncbi.nlm.nih.gov/25052732/
- See also: Follow-up of implant survival comparing ficoll and bone marrow aspirate concentrate methods for hard tissue regeneration with mesenchymal stem cells in humans — http://pubmed.ncbi.nlm.nih.gov/24804168/
- See also: Double Centrifugation Versus Single Centrifugation of Bone Marrow Aspirate Concentrate in Sinus Floor Elevation: A Pilot Study — https://pubmed.ncbi.nlm.nih.gov/26800181/
- See also: Combining autologous bone marrow mononuclear cells seeded on collagen sponge with Nano Hydroxyapatite, and platelet-rich fibrin — https://pubmed.ncbi.nlm.nih.gov/30196860/
- See also: Dimensional ridge alterations following tooth extraction — https://pubmed.ncbi.nlm.nih.gov/15691354/
- See also: Clinical effect of platelet-rich fibrin on the preservation of the alveolar ridge following tooth extraction — https://pubmed.ncbi.nlm.nih.gov/29456635/
- See also: Bone marrow-derived mesenchymal stem cells enhance bone marrow regeneration in dental extraction sockets — https://keio.pure.elsevier.com/en/publications/bone-marrow-derived-mesenchymal-stem-cells-enhance-bone-marrow-re
- See also: A qualitative and quantitative analysis of autologous human multipotent adult stem cells derived from three anatomic areas by marrow aspiration: tibia, anterior ilium, and posterior ilium — https://pubmed.ncbi.nlm.nih.gov/24066346/
- See also: Clinical Outcomes of Socket Preservation Using Bovine-Derived Xenograft Collagen and Collagen Membrane Post-Tooth Extraction — https://pubmed.ncbi.nlm.nih.gov/28817143/
- See also: Xenograft versus extraction alone for ridge preservation after tooth removal — https://pubmed.ncbi.nlm.nih.gov/18672985/